CLINICAL TRIAL: NCT07160127
Title: The Efficacy and Safety of Chinese Herbal Formula TJAOA103 for the Treatment of Genitourinary Syndrome of Menopause: A Prospective and Single-Arm Study
Brief Title: A Clinical Study of Chinese Herbal Formula TJAOA103 in Treating Genitourinary Syndrome of Menopause
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jinjin Zhang, Associate Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202508073-GSM
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Genitourinary Syndrome of Menopause (GSM)
Keywords: Genitourinary Syndrome of Menopause; Traditional Chinise Medicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJAOA103 (Experimental): Once enrolled, participants will be administered TJAOA103 for 4 to 12 weeks.
  Interventions: Drug: TJAOA103

INTERVENTIONS:
Drug: TJAOA103 — Once enrolled, participants will be administered TJAOA103 for 4 to 12 weeks. TJAOA103 should be taken orally twice a day, one sack each time. Dissolve it in about 200 mL of warm water and drink it all. Participants can take it half an hour before breakfast in the morning and half an hour before bedtime in the evening.

SUMMARY:
The goal of this clinical trial is to learn if Chinese herbal formula TJAOA103 works to treat genitourinary syndrome of menopause (GSM). It will also learn about the safety of TJAOA103. The main questions it aims to answer are:

1. Does TJAOA103 alleviate the symptoms of GSM in participants or have any other benefits?
2. What medical problems do participants have when taking TJAOA103? Researchers will conduct a pre-post comparison to see if TJAOA103 works to treat GSM.

Participants will:

1. Take TJAOA103 twice daily for 4 to 12 weeks.
2. Complete the tests and/or questionnaires on schedule through online follow-up or outpatient visits.
3. Record their use of TJAOA103 and any adverse events.

DETAILED DESCRIPTION:
Genitourinary syndrome of menopause (GSM) refers to a collection of symptoms and signs such as atrophy of the genital and urinary tracts and sexual dysfunction in women during the menopausal transition and postmenopausal period due to the decline in estrogen and other sex hormone levels. The primary pathogenesis is rooted in ovarian aging. GSM not only causes persistent discomfort and increases the risk of infections but also significantly impairs sexual function and self-esteem in middle-aged and older women. Furthermore, the failure of ovarian hormone function will markedly elevate the risk of aging-related diseases such as cardiovascular events, Alzheimer's disease, and osteoporosis in these patients, shortening their healthspan and increasing all-cause mortality. Therefore, timely intervention for GSM is crucial.

At present, vaginal moisturizers, lubricants, and vaginal estrogen preparations are commonly used in clinical practice to alleviate the symptoms of GSM. Vaginal moisturizers and lubricants help protect the vaginal epithelium and maintain an acidic vaginal environment, but may cause vaginal burning, infections, or allergic reactions. Vaginal estrogen preparations exert their effects on estrogen receptors within the genitourinary system, yet the long-term safety remains uncertain. Ospemifene, a selective estrogen receptor modulator, is another treatment option; however, its weak estrogenic effects may pose risks of thrombosis or endometrial thickening with prolonged use. In addition, laser therapy has also been employed for GSM, but carries potential safety risks including vaginal burns, scarring, and chronic pain.

Traditional Chinese medicine (TCM) possesses distinctive advantages in anti-aging strategies, addressing both symptoms and root causes with commendable safety profiles, thereby rendering it particularly appropriate for middle-aged and elderly populations. Numerous studies have demonstrated the effectiveness of TCM in the management of GSM-related conditions, such as postmenopausal vaginal dryness, atrophic vaginitis, and menopausal urethral syndrome. However, due to the limited understanding of the disease, existing TCM prescriptions have lacked specificity for GSM and often rely on empirical combinations without solid scientific foundation. To solve this problem, we have invented a novel TCM formula, Tongji Anti-Ovarian Aging 103 (TJAOA103). First, we performed an extensive literature retrieval to collect TCM prescriptions effective in alleviating GSM-associated symptoms. Using the TCM Inheritance Support System and the TCM Systems Pharmacology Database and Analysis Platform, we screened out a variety of candidate Chinese herbs and combinations with potential therapeutic effects on GSM, based on its pathogenesis. Then, a panel of senior experts in gynecology, TCM, and pharmacy thoroughly discussed the pharmacological actions, synergistic effects, contraindications, and dosages of these herbs, and developed the initial formula of TJAOA103. Subsequently, we utilized multiple models to verify the safety and effectiveness of TJAOA103, and further optimized the formulation.

This is a prospective, single-arm clinical study designed to evaluate the safety and efficacy of the TCM formula TJAOA103 in women diagnosed with GSM. Using a pre-post analysis, we will assess the improvements in clinical symptoms, signs, sexual function, genitourinary health, and quality of life in participants with GSM following TJAOA103 administration to provide a safe and reliable novel therapeutic strategy for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 45-70 years during the menopausal transition or postmenopausal period.
2. Presence of at least one moderate-to-severe (score ≥ 2) symptom of GSM, including vulvovaginal dryness, or vulvovaginal itching/irritation, or vulvovaginal burning/pain, or dyspareunia, or dysuria/urinary frequency/urgency.
3. Willing to participate in this trial and sign a written informed consent form.

Exclusion Criteria:

1. Acute or recurrent genitourinary infection.
2. Acute or chronic dermatosis of the vulva or vagina.
3. A grade 3 or higher degree of prolapse according to the Pelvic Organ Prolapse Quantification (POP-Q) system.
4. Unexplained abnormal uterine bleeding.
5. Ovarian/adnexal mass ≥ 4 cm, or adenomyosis, or adenomyoma/uterine myoma ≥ 4 cm.
6. Breast Imaging Reporting and Data System (BI-RADS) classification of breast ultrasound ≥ 4.
7. Presence of precancerous lesions or diagnosed malignancy.
8. Liver or kidney function indicators (ALT, AST, Urea, Cr) exceeding the upper limits of reference ranges upon repeated testing.
9. Severe primary diseases of the nervous, circulatory, respiratory, digestive, urinary or hematopoietic systems; or mental diseases;
10. Known allergy to any specific ingredient of the trial drugs.
11. Systemic hormone therapy within the past 2 months.
12. Application of vaginal moisturizers, lubricants, hormone preparations, or alternative therapies for GSM within the past month.
13. Current participation in another clinical trial or participation in another trial within the past month.
14. Unwillingness to discontinue the use of moisturizers, lubricants, or any form of hormonal drugs during the trial.
15. Other conditions deemed unsuitable for participation by the investigators.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
severity of the most bothersome symptom (MBS) | From enrollment to the end of treatment at 4 or 12 weeks
  The MBS is derived from a selected list of common GSM symptoms, including vulvovaginal dryness, vulvovaginal itching/irritation, vulvovaginal burning/pain, dyspareunia, and dysuria/urinary frequency/urgency. At baseline, participants will be instructed to rate the severity of each symptom as absent (0), mild (1), moderate (2), or severe (3). They will then be asked to select a single MBS among those symptoms they classify as moderate or severe (i.e., a score ≥ 2). The MBS will be tracked through to the end of treatment, and the changes in its severity will be used to assess symptomatic improvement.

SECONDARY OUTCOMES:
total score of GSM symptoms | From enrollment to the end of treatment at 4 or 12 weeks
  The total score, which ranges from 2 to 15, is the sum of the five individual symptom scores. The higher the score, the more severe the GSM symptoms are.
score for a specific GSM symptom | From enrollment to the end of treatment at 4 or 12 weeks
  The self-assessed severity score for a specific GSM symptom is assigned as 0, 1, 2, or 3 points, corresponding respectively to absent, mild, moderate, and severe.
Vaginal Health Index Score (VHIS) | From enrollment to the end of treatment at 4 or 12 weeks
  The total score of VHIS ranges from 5 to 25. The lower the score, the worse the vaginal health condition.
vaginal pH | From enrollment to the end of treatment at 4 or 12 weeks
  A pH level of 4.6 or above indicates vaginal atrophy.
Female Sexual Function Index-6 (FSFI-6) | From enrollment to the end of treatment at 4 or 12 weeks
  The score of FSFI-6 ranges from 2 to 30. A score of 19 or less is considered an indication of female sexual dysfunction.
Overactive Bladder Syndrome Score (OABSS) | From enrollment to the end of treatment at 4 or 12 weeks
  The total OABSS score ranges from 0 to 15. When the score for urinary urgency is 2 or higher, and the total OABSS score is 3 or higher, a diagnosis of overactive bladder syndrome (OAB) can be made. Generally, a total score of 3 to 5 indicates mild OAB, 6 to 11 indicates moderate OAB, and ≥12 indicates severe OAB.
score of International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | From enrollment to the end of treatment at 4 or 12 weeks
  The score of ICIQ-SF ranges from 0 to 21. A higher score indicates more severe urinary incontinence symptoms and a greater impact on the patient's daily life.
score of Menopause-Specific Quality of Life Questionnaire (MENQOL) | From enrollment to the end of treatment at 4 or 12 weeks
  The MENQOL consists of 4 domains, namely vasomotor, psychosocial, physical, and sexual functioning, with a total of 29 items. Participants are instructed to evaluate the existence and degree of bother from their symptoms using a 7-point Likert scale, where higher scores indicate a greater degree of bothersome symptoms. The score for each domain is calculated as the average score of its individual items. The total score is the mean of the four domain scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China